CLINICAL TRIAL: NCT04981782
Title: Passive Cervical Range of Motion in Infants With and Without Torticollis, Before, During and After Chiropractic Treatment
Brief Title: Passive Cervical Range of Motion in Infants
Acronym: CROMinfants
Status: Completed | Type: Observational
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-02328
Record Dates: First submitted 2021-07-20; First posted 2021-07-29 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Arthrogenic Torticollis
Keywords: arthrogenic Torticollis; cervical range of motion; infant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthy subjects: No intervention
  Infants will be measured at different time points. At the age of 3,4,6 and 9 months.
  Interventions: Other: No study specific intervention, regular care.
- torticollis group: No intervention
  Infants will be measured at their visit to a Chiropractor. Before and after treatment.
  Interventions: Other: No study specific intervention, regular care.

INTERVENTIONS:
Other: No study specific intervention, regular care. — Chiropractic care (regular care)
  Other Names: chiropractic treatment

SUMMARY:
Infants with and without torticollis will be measured at different time points to assess their passive cervical spine range of motion (pCROM).

DETAILED DESCRIPTION:
Infants at the age of 2 to 12 month will be measured at several time points to assess their passive cervical range of motion. One group will include healthy subjects, the other group infants with a diagnosed torticollis. Healthy subjects will be measured at the age of 3, 4, 6 and 9 months. Infants diagnosed with torticollis, at their visit at a Chiropractor and one week later.

ELIGIBILITY:
Inclusion Criteria:

* age 2-12 month
* signed informed consent
* diagnosed with torticollis

Exclusion Criteria:

* defense reaction e.g. crying, screaming
* other illnesses
* neck trauma
* neck surgery
* developmental delay

Ages: 2 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: infants with torticollis
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
passive cervical range of motion (pCROM) | baseline
  The ability of passive movement of the cervical spine will be assessed
passive cervical range of motion (pCROM) | three months
  The ability of passive movement of the cervical spine will be assessed
passive cervical range of motion (pCROM) | six months
  The ability of passive movement of the cervical spine will be assessed
passive cervical range of motion (pCROM) | four months
  The ability of passive movement of the cervical spine will be assessed
passive cervical range of motion (pCROM) | nine months
  The ability of passive movement of the cervical spine will be assessed

SECONDARY OUTCOMES:
Demographic data child | baseline
  specific data of the child is gathered
Demographic data mother | baseline
  specific data of the mother is collected

CONTACTS AND LOCATIONS:
Overall Officials: Petra Schweinhardt, PhD, Study Chair — University of Zurich and Balgrist University Hospital
Locations (2):
- Switzerland (2):
  - Balgrist University Hospital, Zurich, Canton of Zurich
  - Balgrist University Hospital, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Langenfeld A, Paravicini I, Hobaek Siegenthaler M, Wehrli M, Hausler M, Bergander T, Schweinhardt P. Subjective and Objective Assessment of the Preferred Rotational Cervical Spine Position in Infants with an Upper Cervical Spine Dysfunction: A Cross-Sectional Study. Children (Basel). 2024 Dec 13;11(12):1515. doi: 10.3390/children11121515. PMID 39767944